CLINICAL TRIAL: NCT00002492
Title: CLINICAL AND PHARMACOLOGICAL STUDY OF CHEMOTHERAPY IN SOFT TISSUE SARCOMA
Brief Title: Combination Chemotherapy in Treating Patients With Soft Tissue Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Miami (Other)
Purpose: Treatment
Other Study IDs: 89253; SCCC-1989032 (Other: University of Miami Sylvester Comprehensive Cancer Center); NCI-V92-0066
Record Dates: First submitted 1999-11-01; First posted 2004-04-22 (Estimated); Last update posted 2016-12-15 (Estimated); Status verified 2016-12

CONDITIONS: Sarcoma
Keywords: stage I adult soft tissue sarcoma; stage II adult soft tissue sarcoma; stage III adult soft tissue sarcoma
MeSH Terms: conditions — Sarcoma | interventions — Cisplatin; Doxorubicin; Brachytherapy; Radiotherapy

INTERVENTIONS:
Drug: cisplatin
Drug: doxorubicin hydrochloride
Drug: isolated limb perfusion
Procedure: conventional surgery
Radiation: brachytherapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining cisplatin and doxorubicin in treating patients who have soft tissue sarcoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the response in patients with resectable soft tissue sarcoma of the extremity treated with neoadjuvant intra-arterial cisplatin and IV doxorubicin followed by limb-sparing procedure or amputation, adjuvant IV cisplatin and IV doxorubicin, and radiotherapy. II. Determine the chemotherapeutic response in tumor specimens of patients treated with this regimen.

OUTLINE: Neoadjuvant chemotherapy: Patients undergo arterial cannulation followed by cisplatin intra-arterially over 4 hours on day 1 and doxorubicin IV (beginning 15 minutes after completion of cisplatin infusion) on days 1-3. Treatment continues every 3 weeks for 2 courses in the absence of unacceptable toxicity. Patients undergo amputation or limb-sparing wide excision, as feasible, approximately 4 weeks after the second course. If surgery cannot be scheduled at this time for logistical reasons, a third course may be administered. Patients with an estimated tumor kill of at least 50% receive adjuvant chemotherapy as outlined below. Patients undergoing limb-sparing wide excision receive post-operative radiotherapy as outlined below. Adjuvant chemotherapy: Beginning 3-4 weeks after surgery, patients receive cisplatin IV over 4 hours on day 1 and doxorubicin as above on days 1-3. Treatment continues every 3 weeks for 4 courses in the absence of disease progression, stable disease, or unacceptable toxicity. Patients undergoing radiotherapy receive the final 3 courses of chemotherapy after completion of radiotherapy. Post-operative radiotherapy: Beginning after the first postoperative chemotherapy course and within 8 weeks after surgery, patients receive radiotherapy 5 days a week for 7-8 weeks. An interstitial implant using iridium Ir 192 may be used to administer the final doses of radiotherapy.

PROJECTED ACCRUAL: A total of 40 patients will be accrued for this study within 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Diagnosis of intermediate- or high-grade soft tissue sarcoma of the extremity amenable to limb-sparing procedure or amputation Buttocks or shoulder lesions allowed if an artery is available for cannulation No metastasis

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Not specified Life expectancy: Not specified Hematopoietic: WBC at least 3,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin less than 2.0 mg/dL Renal: Creatinine clearance at least 60 mL/min Cardiovascular: Ejection fraction at least 50% by MUGA scan No history of congestive heart failure or severe angina pectoris Other: No other prior malignancy except basal cell skin cancer or carcinoma in situ of the cervix Not pregnant Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy Endocrine therapy: Not specified Radiotherapy: No prior radiotherapy Surgery: See Disease Characteristics

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1991-11; Primary Completion 2000-02 (Actual); Study Completion 2000-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pasquale W. Benedetto, MD, Study Chair — University of Miami Sylvester Comprehensive Cancer Center
Locations (1):
- Sylvester Cancer Center, University of Miami, Miami, Florida, United States